CLINICAL TRIAL: NCT02667353
Title: Structural Brain Plasticity in Elderly Depressed Patients Following Electroconvulsive Therapy
Brief Title: Neurorestorative Effects of Electroconvulsive Therapy (ECT) in Patients With Severe Late Life Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: VU University of Amsterdam (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: S53144
Record Dates: First submitted 2016-01-18; First posted 2016-01-28 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Depression
Keywords: electroconvulsive; hippocampus; elderly; working mechanism
MeSH Terms: conditions — Depression | interventions — Electroconvulsive Therapy; Etomidate; Anesthetics; Succinylcholine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- electroconvulsive therapy (Other): only one arm in this study: patients who are treated with electroconvulsive therapy and have been given anesthesia with etomidate and succinylcholine
  Interventions: Procedure: ECT; Drug: Etomidate; Drug: Succinylcholine

INTERVENTIONS:
Procedure: ECT — ECT was administered twice a week with a constant-current brief-pulse device (Thymatron, System IV). Motor and electroencephalographic seizures were monitored to ensure adequate duration and quality. Subjects were all treated with right unilateral (RUL) ECT with stimulus intensity 6 times the initial seizure threshold (ST), as determined by empirical dose titration at the first treatment, until remission (Montgomery-Åsberg Depression Rating Scale (MADRS) (27) < 10 in two consecutive ratings with a week interval). Subjects who failed to respond right unilateral ECT after the sixth treatment were switched to bitemporal ECT (1.5x seizure threshold).
  Other Names: electroconvulsive therapy
Drug: Etomidate — Anesthesia was achieved with intravenous administration of etomidate (0.2mg/kg).
  Other Names: anesthetic
Drug: Succinylcholine — Anesthesia was achieved with intravenous administration of succinylcholine (1mg/kg).
  Other Names: muscle relaxant

SUMMARY:
To study the potential neurorestorative effects of electroconvulsive therapy (ECT) in depressed patients by measuring brain derived neurotrophic factor (BDNF) serum levels and hippocampal volumes in severely depressed patients receiving ECT.

DETAILED DESCRIPTION:
The investigators want to study the potential neurorestorative effects of electroconvulsive therapy (ECT) in depressed patients by measuring brain derived neurotrophic factor (BDNF) serum levels and hippocampal volumes in severely depressed patients receiving ECT.

Clinical studies in severely depressed patients have shown that antidepressants and ECT can increase Brain Derived Neurotrophic Factor (BDNF) serum levels. BDNF serum levels will be measured before, during and after ECT. In animal studies this increase in serum BDNF was shown to induce hippocampal mossy fiber sprouting and the investigators want to study this phenomenon in humans. Recently, a volumetric magnetic resonance imaging study showed increased hippocampal volume in patients with depression. Hippocampal volumes will be determined with magnetic resonance imaging scannings including voxel based morphometry. Severe depression is accompanied by a dysfunction of the hypothalamus pituitary adrenal (HPA) axis. Cortisol and several other hormones have psychotropic effects, and their excesses or deficiencies induce states of mania or depression. High levels of cortisol suppress hippocampal neurogenesis. Animal models have shown that this suppressive effect of cortisol on hippocampal neurogenesis could be reversed to normal levels by electroconvulsive stimulation, the animal model for ECT. This animal study is in good accordance with clinical findings.

The investigators hypothesize the following: Increase of brain-derived neurotrophic factor serum levels induced by electroconvulsive therapy are associated with remission and is correlated with a neurorestorative effect, which is an increase of hippocampal volume. Non- response to ECT is explained by either low BDNF serum levels regardless of hippocampus size, or by (more advanced) medial temporal lobe atrophy (beyond a point of no return) despite increased BDNF serum levels.

Additionally, four relevant functional candidate genes will be examined, based on their putative role in neurotrophic processes and/or in treatment response in depression: the brain derived neurotrophic factor gene, the serotonin transporter gene, the vascular endothelial growth factor gene and the apolipoprotein gene.

The investigators will also evaluate cognitive and psychomotor changes following electroconvulsive therapy given their clinical relevance in late life depression.

ELIGIBILITY:
Inclusion Criteria:

* Patients are considered suitable after they were diagnosed as having severe depression according to Diagnostic and Statistical Manual IV (DSM-IV criteria) and were above 55 years of age.

Exclusion Criteria:

* another major psychiatric illness, (a history of) a major neurological illness (including Parkinson's disease, stroke, and dementia) and metal implants precluding Magnetic Resonance Imaging (MRI).

Subjects were included at the University Psychiatric Center Katholieke Universiteit Leuven (KU Leuven), Belgium and Geestelijke Gezondheidszorg in Geest (GGZinGeest), Amsterdam, the Netherlands. The project is part of the project Mood Disorders in Elderly and Electroconvulsive therapy (MODECT).

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2011-06; Primary Completion 2014-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
change in hippocampal volume as assessed by manual delineation following an initial automatic segmentation | 6 months
  Hippocampal volumes were normalized using the following equation: normalised hippocampal volume = original hippocampal volume - linear regression coefficient x (total intracranial volume - mean total intracranial volume). The coefficient was derived from a linear regression of total intracranial volume and original hippocampal volume. Total intracranial volume was obtained from an automated segmentation of grey matter, white matter and cerebrospinal fluid. Intra-rater reliability was determined using randomly selected scans segmented at two time-points at least one month apart. The intra-class correlation coefficient (Cronbach's alfa) was 0.96 for the left hippocampus and 0.95 for the right hippocampus.
change in brain derived neurotrophic factor as assessed by the Emax Immuno Assay system | 4 weeks
  Blood samples were taken between 07:30 am and 09:30 am after an overnight fast. Serum was immediately separated and stored at -85 °celcius until assayed. BDNF protein levels were measured using the Emax Immuno Assay system from Promega according to the manufacturer's protocol (Madison, United States of America), in one laboratory (Maastricht University). Undiluted serum was acid treated as this reliably increased the detectable BDNF in a dilution-dependent way. Greiner Bio-One high affinity 96-well plates were used. Serum samples were diluted 100 times, and the absorbency was read in duplicate using a Bio-Rad (Hercules, United States of America) Benchmark microplate reader at 450 nm.
change of mood as assessed by the Montgomery-Åsberg Depression Rating Scale (MADRS) | up to 1 year
  The MADRS is a ten-item diagnostic questionnaire which psychiatrists use to measure the severity of depressive episodes in patients with mood disorders. Higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60. The questionnaire includes questions on the following symptoms: apparent sadness; reported sadness; inner tension; reduced sleep; reduced appetite; concentration difficulties; lassitude; inability to feel; pessimistic thoughts; suicidal thoughts.

SECONDARY OUTCOMES:
change of cognition as assessed by the mini mental state examination | up to 1 year
  The mini-mental state examination is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment. The test includes questions in a number of areas: the time and place, repeating lists of words, arithmetic, and basic motor skills.
change of psychomotor symptoms as assessed by the CORE (not an acronym) | up to 1 year
  The CORE (this is not an acronym) was used to assess psychomotor symptoms in detail and comprises 18 observable features which are rated on a four-point scale. Summing subsets of the items produces scores on three dimensions found to underlay psychomotor change: non-interactiveness, retardation and agitation.

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu Vandenbulcke, MD PhD, Study Director — Universitaire Ziekenhuizen KU Leuven

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bolwig TG. How does electroconvulsive therapy work? Theories on its mechanism. Can J Psychiatry. 2011 Jan;56(1):13-8. doi: 10.1177/070674371105600104. PMID 21324238
- [Background] Bocchio-Chiavetto L, Zanardini R, Bortolomasi M, Abate M, Segala M, Giacopuzzi M, Riva MA, Marchina E, Pasqualetti P, Perez J, Gennarelli M. Electroconvulsive Therapy (ECT) increases serum Brain Derived Neurotrophic Factor (BDNF) in drug resistant depressed patients. Eur Neuropsychopharmacol. 2006 Dec;16(8):620-4. doi: 10.1016/j.euroneuro.2006.04.010. Epub 2006 Jun 6. PMID 16757154
- [Background] Bolwig TG, Madsen TM. Electroconvulsive therapy in melancholia: the role of hippocampal neurogenesis. Acta Psychiatr Scand Suppl. 2007;(433):130-5. doi: 10.1111/j.1600-0447.2007.00971.x. PMID 17280579
- [Background] Chen AC, Shin KH, Duman RS, Sanacora G. ECS-Induced mossy fiber sprouting and BDNF expression are attenuated by ketamine pretreatment. J ECT. 2001 Mar;17(1):27-32. doi: 10.1097/00124509-200103000-00006. PMID 11281511
- [Background] Duman RS, Monteggia LM. A neurotrophic model for stress-related mood disorders. Biol Psychiatry. 2006 Jun 15;59(12):1116-27. doi: 10.1016/j.biopsych.2006.02.013. Epub 2006 Apr 21. PMID 16631126
- [Background] Egan MF, Kojima M, Callicott JH, Goldberg TE, Kolachana BS, Bertolino A, Zaitsev E, Gold B, Goldman D, Dean M, Lu B, Weinberger DR. The BDNF val66met polymorphism affects activity-dependent secretion of BDNF and human memory and hippocampal function. Cell. 2003 Jan 24;112(2):257-69. doi: 10.1016/s0092-8674(03)00035-7. PMID 12553913
- [Background] Fisman M, Rabheru K, Hegele RA, Sharma V, Fisman D, Doering M, Appell J. Apolipoprotein E polymorphism and response to electroconvulsive therapy. J ECT. 2001 Mar;17(1):11-4. doi: 10.1097/00124509-200103000-00003. PMID 11281508
- [Background] Marano CM, Phatak P, Vemulapalli UR, Sasan A, Nalbandyan MR, Ramanujam S, Soekadar S, Demosthenous M, Regenold WT. Increased plasma concentration of brain-derived neurotrophic factor with electroconvulsive therapy: a pilot study in patients with major depression. J Clin Psychiatry. 2007 Apr;68(4):512-7. doi: 10.4088/jcp.v68n0404. PMID 17474805
- [Background] Montgomery SA, Asberg M. A new depression scale designed to be sensitive to change. Br J Psychiatry. 1979 Apr;134:382-9. doi: 10.1192/bjp.134.4.382. PMID 444788
- [Background] Newton SS, Collier EF, Hunsberger J, Adams D, Terwilliger R, Selvanayagam E, Duman RS. Gene profile of electroconvulsive seizures: induction of neurotrophic and angiogenic factors. J Neurosci. 2003 Nov 26;23(34):10841-51. doi: 10.1523/JNEUROSCI.23-34-10841.2003. PMID 14645477
- [Background] Nordanskog P, Dahlstrand U, Larsson MR, Larsson EM, Knutsson L, Johanson A. Increase in hippocampal volume after electroconvulsive therapy in patients with depression: a volumetric magnetic resonance imaging study. J ECT. 2010 Mar;26(1):62-7. doi: 10.1097/YCT.0b013e3181a95da8. PMID 20190603
- [Background] Oudega ML, van Exel E, Wattjes MP, Comijs HC, Scheltens P, Barkhof F, Eikelenboom P, de Craen AJ, Beekman AT, Stek ML. White matter hyperintensities, medial temporal lobe atrophy, cortical atrophy, and response to electroconvulsive therapy in severely depressed elderly patients. J Clin Psychiatry. 2011 Jan;72(1):104-12. doi: 10.4088/JCP.08m04989blu. Epub 2010 Aug 24. PMID 20816035
- [Background] Sapolsky RM. Depression, antidepressants, and the shrinking hippocampus. Proc Natl Acad Sci U S A. 2001 Oct 23;98(22):12320-2. doi: 10.1073/pnas.231475998. No abstract available. PMID 11675480
- [Background] Segi-Nishida E, Warner-Schmidt JL, Duman RS. Electroconvulsive seizure and VEGF increase the proliferation of neural stem-like cells in rat hippocampus. Proc Natl Acad Sci U S A. 2008 Aug 12;105(32):11352-7. doi: 10.1073/pnas.0710858105. Epub 2008 Aug 5. PMID 18682560
- [Background] Steffens DC, Byrum CE, McQuoid DR, Greenberg DL, Payne ME, Blitchington TF, MacFall JR, Krishnan KR. Hippocampal volume in geriatric depression. Biol Psychiatry. 2000 Aug 15;48(4):301-9. doi: 10.1016/s0006-3223(00)00829-5. PMID 10960161
- [Background] UK ECT Review Group. Efficacy and safety of electroconvulsive therapy in depressive disorders: a systematic review and meta-analysis. Lancet. 2003 Mar 8;361(9360):799-808. doi: 10.1016/S0140-6736(03)12705-5. PMID 12642045
- [Background] Vaidya VA, Siuciak JA, Du F, Duman RS. Hippocampal mossy fiber sprouting induced by chronic electroconvulsive seizures. Neuroscience. 1999 Mar;89(1):157-66. doi: 10.1016/s0306-4522(98)00289-9. PMID 10051225
- [Derived] Wagenmakers MJ, Oudega ML, Klaus F, Wing D, Orav G, Han LKM, Binnewies J, Beekman ATF, Veltman DJ, Rhebergen D, van Exel E, Eyler LT, Dols A. BrainAge of patients with severe late-life depression referred for electroconvulsive therapy. J Affect Disord. 2023 Jun 1;330:1-6. doi: 10.1016/j.jad.2023.02.047. Epub 2023 Feb 27. PMID 36858270
- [Derived] Wagenmakers MJ, Oudega ML, Bouckaert F, Rhebergen D, Beekman ATF, Veltman DJ, Sienaert P, van Exel E, Dols A. Remission Rates Following Electroconvulsive Therapy and Relation to Index Episode Duration in Patients With Psychotic Versus Nonpsychotic Late-Life Depression. J Clin Psychiatry. 2022 Aug 10;83(5):21m14287. doi: 10.4088/JCP.21m14287. PMID 35950901
- [Derived] Carlier A, Rhebergen D, Veerhuis R, Schouws S, Oudega ML, Eikelenboom P, Bouckaert F, Sienaert P, Obbels J, Stek ML, van Exel E, Dols A. Inflammation and Cognitive Functioning in Depressed Older Adults Treated With Electroconvulsive Therapy: A Prospective Cohort Study. J Clin Psychiatry. 2021 Aug 10;82(5):20m13631. doi: 10.4088/JCP.20m13631. PMID 34383393